CLINICAL TRIAL: NCT00542295
Title: Efficacy and Safety of Meteospasmyl® in Irritable Bowel Syndrome. a 4-Week, Multicentre, Double-Blind, Randomised, Placebo-Controlled Phase IV Trial
Brief Title: Efficacy and Safety of Meteospasmyl® in Irritable Bowel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires Mayoly Spindler (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMTO601
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2008-09

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — alverine; Simethicone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: alverine citrate and simeticone
- B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: alverine citrate and simeticone
  Other Names: Meteospasmyl®
  Arms: A
Drug: placebo
  Arms: B

SUMMARY:
To assess the effectiveness of alverine citrate and simeticone on IBS symptoms according to the latest recommended design

ELIGIBILITY:
Inclusion Criteria:

* male or female ambulatory patients, aged 18-75 years
* with IBS as defined by Rome III criteria

Exclusion Criteria:

* Functional bowel disorder other than IBS,
* Underlying cause for symptomatology, which excludes IBS diagnosis,
* Gastro-intestinal cancer or significant gastro-intestinal surgical background,
* Any acute/uncontrolled systemic pathology

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Subject self assessment of abdominal pain/discomfort | Baseline and 4 weeks

SECONDARY OUTCOMES:
IBS life impact, overall treatment assessment, concomitant factors | Baseline and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Ducrotte, M.D, Study Chair
Locations (13):
- Hungary (8):
  - Budapest
  - Debrecen
  - Győr
  - Gyula
  - Miskolc
  - Siofolk
  - Szeged
  - Székesfehérvár
- Poland (5):
  - Bydgoszcz
  - Katowice
  - Oława
  - Szczecin
  - Wroclaw